CLINICAL TRIAL: NCT01666652
Title: A Phase I, Randomized, Placebo-Controlled, Observer-blind, Two-dose (0-28 Day Schedule) Primary Vaccination Study of Walter Reed Army Institute of Research (WRAIR) Tetravalent Dengue Virus Purified Inactivated Vaccine (TDENV-PIV) in Healthy Adults in a Non-Endemic Region
Brief Title: A Two-dose Primary Vaccination Study of a Tetravalent Dengue Virus Purified Inactivated Vaccine vs. Placebo in Healthy Adults
Acronym: DPIV-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-11-23; WRAIR 1923 (Other: WRAIR); GSK 116289 (Other: GlaxoSmithKline (GSK)); A-17355.b (Other: USAMRMC HRPO)
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Dengue Fever
Keywords: Dengue; Dengue fever; Dengue Hemorrhagic Fever; Flavivirus
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TDENV-PIV alum4 (Experimental): 4 µg TDENV-PIV with Alum adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: 4 µg TDENV-PIV with Alum adjuvant
- TDENV-PIV AS01E1 (Experimental): 1 µg TDENV-PIV with AS01E1 adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: 1 µg TDENV-PIV with AS01E1 adjuvant
- TDENV-PIV AS03B1 (Experimental): 1 µg TDENV-PIV with AS03B1 adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: 1 µg TDENV-PIV with AS03B1 adjuvant
- Placebo (Placebo Comparator): Phosphate buffered saline; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Other: Phosphate buffered saline
- TDENV-PIV alum1 (Experimental): 1 µg TDENV-PIV with Alum adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: 1 µg TDENV-PIV with Alum adjuvant

INTERVENTIONS:
Biological: 4 µg TDENV-PIV with Alum adjuvant
  Arms: TDENV-PIV alum4
Biological: 1 µg TDENV-PIV with AS03B1 adjuvant
  Arms: TDENV-PIV AS03B1
Other: Phosphate buffered saline
  Arms: Placebo
Biological: 1 µg TDENV-PIV with Alum adjuvant
  Arms: TDENV-PIV alum1
Biological: 1 µg TDENV-PIV with AS01E1 adjuvant
  Arms: TDENV-PIV AS01E1

SUMMARY:
The study is designed to afford a safety and immunogenicity assessment of three Tetravalent Dengue Virus-Purified Inactivated Vaccine(TDENV-PIV) vaccine candidates.

DETAILED DESCRIPTION:
The study is designed to afford a safety and immunogenicity assessment of three Tetravalent Dengue Virus-Purified Inactivated Vaccine(TDENV-PIV) vaccine candidates, each formulated with a different adjuvant: either aluminum hydroxide, AS01E or AS03B (adjuvants used in Glaxo Smith Kline (GSK) Biologicals' hepatitis B candidate vaccine, malaria candidate vaccine and pandemic flu vaccine, respectively). Each vaccine candidate will contain 1 µg of purified virus antigen per each of the four DENV types. Additionally, the study will evaluate an alum adjuvanted TDENV-PIV vaccine candidate containing 4 µg of purified virus antigen per each of the four DENV types. The control group will receive a saline placebo. All experimental vaccinations will be administered according to a 2-dose schedule, 28 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits, etc.)
* A male or female between 18 and 39 years of age (inclusive) at the time of consent
* Written informed consent obtained from the subject
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Female subjects of non-childbearing potential (non-childbearing potential is defined as having either a current tubal ligation at least three months prior to enrollment, hysterectomy, ovariectomy, or is post-menopause). See Definition of Terms for adequate contraception.
* Female subjects of childbearing potential may be enrolled in the study, if the subject has:

  * Practiced adequate contraception for 30 days prior to vaccination, and
  * A negative urine pregnancy test on the day of vaccination, and
  * Agreed to continue adequate contraception until two months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines/placebo during the period starting 30 days preceding the first dose of study vaccine/placebo and/or planned use during the study period
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to the first vaccine/placebo dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent; inhaled and topical steroids are allowed)
* Planned administration or administration of a vaccine/product not foreseen by the study protocol during the period starting 30 days prior to the first dose of vaccine/placebo until after the visit at Day 56 (if influenza activity warrants vaccination of healthy young adults, influenza vaccination will be encouraged and will not lead to study exclusion)
* Planned administration of any flavivirus vaccine for the entire study duration
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency
* History of, or current auto-immune disease
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/placebo or related to a study procedure
* Major congenital defects or serious chronic illness
* History of any neurological disorders or seizures
* Acute disease and/or fever (≥37.5°C/99.5°F oral body temperature) at the time of enrollment (a subject with a minor illness, i.e., mild diarrhea, mild upper respiratory infection, etc., without fever, may be enrolled at the discretion of the investigator)
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality,as determined by physical examination or laboratory screening tests
* Administration of immunoglobulins and/or any blood products during the period starting 90 days preceding the first dose of study vaccine/placebo or planned administration during the study period
* History of chronic alcohol consumption and/or drug abuse
* Pregnant or lactating female or female planning to become pregnant or planning to discontinue contraceptive precautions
* A planned move to a location that will prohibit participating in the trial until study end for the participant
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Subject seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
* Safety laboratory test results that are outside the acceptable values at screening. The following values are not acceptable:

  * >110% upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, creatinine, serum urea nitrogen (SUN) and bilirubin (total and direct)
  * <100% lower limit of normal (LLN) or > 120% ULN for hemoglobin, hematocrit and platelet count
  * <75% LLN or >110% ULN for total white blood cell count (WBC) Note that all screening laboratory results must be either within normal limits (WNL) or no more than Grade l not clinically significant (NCS)

(LLN=lower limit of normal; ULN= upper limit of normal, WNL= within normal limits, NCS= not clinically significant)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leyi Lin, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- WRAIR, Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schmidt AC, Lin L, Martinez LJ, Ruck RC, Eckels KH, Collard A, De La Barrera R, Paolino KM, Toussaint JF, Lepine E, Innis BL, Jarman RG, Thomas SJ. Phase 1 Randomized Study of a Tetravalent Dengue Purified Inactivated Vaccine in Healthy Adults in the United States. Am J Trop Med Hyg. 2017 Jun;96(6):1325-1337. doi: 10.4269/ajtmh.16-0634. PMID 28719287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled healthy male and non-pregnant, non-breast-feeding, female subjects between the ages of 18 and 39 (inclusive). Subjects were enrolled at the CTC, WRAIR, Silver Spring, Maryland, US. Subjects were not screened for prior flavivirus infection.
Groups:
- TDENV-PIV alum1: 1 µg TDENV-PIV with Alum adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  1 µg TDENV-PIV with Alum adjuvant
- TDENV-PIV alum4: 4 µg TDENV-PIV with Alum adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  4 µg TDENV-PIV with Alum adjuvant
- TDENV-PIV AS01E1: 1 µg TDENV-PIV with AS01E1 adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  1 µg TDENV-PIV with AS01E1 adjuvant
- TDENV-PIV AS03B1: 1 µg TDENV-PIV with AS03B1 adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  1 µg TDENV-PIV with AS03B1 adjuvant
- Placebo: Phosphate buffered saline; 0.5 mL intramuscular injection at 0 and 28 days
  Phosphate buffered saline
Period: Overall Study
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Started | 20 | 20 | 20 | 20 | 20
Completed | 18 | 19 | 19 | 16 | 19
Not Completed | 2 | 1 | 1 | 4 | 1
Not completed — Serious Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Moved from study area | 1 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (5.68) | 26.1 (4.55) | 28.0 (6.86) | 28.4 (5.56) | 28.3 (5.47) | 27.8 (5.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 7 | 11 | 7 | 43
  Male | 9 | 13 | 13 | 9 | 13 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 1 | 0 | 1 | 2
  Asian-Central/South Asian | 0 | 1 | 1 | 2 | 0 | 4
  Asian-East Asian | 1 | 0 | 0 | 0 | 0 | 1
  White-Caucasian/European | 10 | 4 | 4 | 8 | 8 | 34
  Other | 1 | 2 | 2 | 1 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 20 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events Within the 28 Day Follow-up
Description: Number of subjects with adverse events occurring within days 0-28 following vaccination
Time Frame: Days 0-28
Measure: Count of Participants; unit: Participants
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Participants
  Subjects with any AEs | 10 | 9 | 10 | 14 | 15
  Upper respiratory tract infection | 0 | 2 | 0 | 3 | 0
  Nasopharyngitis | 2 | 0 | 0 | 2 | 2
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 3
  Bradycardia | 0 | 0 | 0 | 0 | 2
  Chills | 0 | 0 | 2 | 0 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 2
  White blood cell count increased | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Incidence of Any Symptoms (Solicited and Unsolicited) Reported During the 7-day Post Vaccination Period. Total Vaccinated Cohort (TVC)
Description: Overall incidence of any symptoms (solicited and unsolicited) reported during the 7-day (days 0-6) post vaccination period in TVC population
Time Frame: Days 0-6 post vaccination
Measure: Number; unit: AEs
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 18 | 19 | 20 | 20
AEs
  Dose 1 | 8 | 12 | 15 | 20 | 13
  Dose 2 | 7 | 9 | 15 | 15 | 11

3. Primary Outcome: Incidence of General Symptoms (Solicited and Unsolicited) Reported During the 7-day Post Vaccination Period, Total Vaccinated Cohort (TVC)
Description: Incidence of General Symptoms (Solicited and Unsolicited) Reported during the 7-day Post Vaccination Period for TVC population. General symptoms are described as fatigue, gastrointestinal symptoms, headache, joint pain, muscle aches and increased temperature (oral).
Time Frame: Days 0-6 post vaccination
Measure: Number; unit: AEs
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 18 | 19 | 20 | 20
AEs
  Dose 1 | 8 | 10 | 12 | 14 | 12
  Dose 2 | 2 | 7 | 10 | 14 | 11

4. Primary Outcome: Incidence of Local Symptoms (Solicited and Unsolicited) Reported During the 7-day Post Vaccination Period, Total Vaccinated Cohort (TVC)
Description: Incidence of Local Symptoms (Solicited and Unsolicited) Reported during the 7-day Post Vaccination Period in TVC population. Local symptoms are described as pain, redness and swelling.
Time Frame: Days 0-6 post vaccination
Measure: Number; unit: AEs
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 18 | 19 | 20 | 20
AEs
  Dose 1 | 6 | 7 | 15 | 17 | 2
  Dose 2 | 5 | 6 | 14 | 12 | 2

5. Primary Outcome: Summary of Subjects With Serious Adverse Events
Description: Summary of subjects with serious adverse events through out the study
Time Frame: days 0-392
Measure: Count of Participants; unit: Participants
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Participants
  Asthma | 0 | 0 | 1 | 0 | 0
  Miscarriage | 0 | 0 | 0 | 1 | 0
  Worsening abdominla discomfort | 0 | 0 | 0 | 1 | 0
  Gunshot wound | 0 | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Subjects With Laboratory Values Within and Outside the Normal Ranges and With Different Grade of Adverse Event From Screening to Day 56 Visit
Description: The percentage of subjects with hematological and biochemical laboratory values within and outside the normal ranges and with different grade of AE were tabulated with exact 95% CI at baseline and at each specified timepoint. Safety laboratory assays were performed at a WRAIR-designated Clinical Laboratory Improvement Amendments-certified laboratory. All safety-related clinical laboratory values were reviewed and all abnormal values were assessed by the investigators as clinically significant or not, with respect to safety.
  PRE = Pre-vaccination, Day 0 visit PI(D7) = Post-dose 1, Day 7 visit PI(D28) = Post-dose 1, Day 28 visit PII(D35) = Post-dose 2, Day 35 visit PII(D56) = Post-dose 2, Day 56 visit PII(M4) = Post-dose 2, Month 4 visit PII(M7) = Post-dose 2, Month 7 visit PII(M10) = Post-dose 2, Month 10 visit PII(M13) = Post-dose 2, Month 13 visit
Time Frame: day 56 visit
Measure: Count of Participants; unit: Participants
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Participants
  ALAT: SCR: Below LLN | 0 | 0 | 0 | 1 | 1
  ALAT: SCR: Normal | 20 | 20 | 20 | 19 | 19
  ALAT: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  ALAT: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  ALAT: SCR: Missing | 0 | 0 | 0 | 0 | 0
  ALAT: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ALAT: PRE: Below LLN | 0 | 0 | 1 | 1 | 0
  ALAT: PRE: Normal | 19 | 19 | 19 | 19 | 20
  ALAT: PRE: Grade 1-2 | 1 | 1 | 0 | 0 | 0
  ALAT: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  ALAT: PRE: Missing | 0 | 0 | 0 | 0 | 0
  ALAT: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ALAT: PI(D7): Below LLN | 0 | 1 | 1 | 2 | 1
  ALAT: PI(D7): Normal | 20 | 18 | 19 | 18 | 19
  ALAT: PI(D7): Grade 1-2 | 0 | 1 | 0 | 0 | 0
  ALAT: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  ALAT: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  ALAT: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ALAT: PI(D28): Below LLN | 0 | 0 | 0 | 2 | 0
  ALAT: PI(D28): Normal | 20 | 19 | 20 | 17 | 20
  ALAT: PI(D28): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  ALAT: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  ALAT: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  ALAT: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ALAT: PII(D35): Below LLN | 0 | 0 | 0 | 1 | 1
  ALAT: PII(D35): Normal | 20 | 18 | 19 | 18 | 19
  ALAT: PII(D35): Grade 1-2 | 0 | 1 | 1 | 0 | 0
  ALAT: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  ALAT: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  ALAT: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ALAT: PII(D56): Below LLN | 0 | 0 | 0 | 1 | 1
  ALAT: PII(D56): Normal | 19 | 19 | 20 | 18 | 19
  ALAT: PII(D56): Grade 1-2 | 1 | 00 | 0 | 0 | 0
  ALAT: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  ALAT: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  ALAT: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  AP: SCR: Below LLN | 0 | 0 | 0 | 1 | 0
  AP: SCR: Normal | 20 | 20 | 20 | 19 | 20
  AP: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  AP: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  AP: SCR: Missing | 0 | 0 | 0 | 0 | 0
  AP: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  AP: PRE: Below LLN | 0 | 0 | 0 | 1 | 0
  AP: PRE: Normal | 20 | 20 | 20 | 19 | 20
  AP: PRE: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  AP: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  AP: PRE: Missing | 0 | 0 | 0 | 0 | 0
  AP: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  AP: PI(D7): Below LLN | 0 | 0 | 0 | 1 | 0
  AP: PI(D7): Normal | 20 | 20 | 20 | 19 | 20
  AP: PI(D7): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  AP: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  AP: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  AP: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  AP: PI(D28): Below LLN | 1 | 0 | 0 | 1 | 0
  AP: PI(D28): Normal | 19 | 19 | 20 | 18 | 20
  AP: PI(D28): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  AP: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  AP: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  AP: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  AP: PII(D35): Below LLN | 1 | 0 | 0 | 1 | 0
  AP: PII(D35): Normal | 19 | 19 | 20 | 18 | 20
  AP: PII(D35): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  AP: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  AP: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  AP: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  AP: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  AP: PII(D56): Normal | 20 | 19 | 20 | 19 | 20
  AP: PII(D56): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  AP: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  AP: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  AP: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ASAT: SCR: Below LLN | 0 | 0 | 0 | 0 | 1
  ASAT: SCR: Normal | 20 | 20 | 20 | 20 | 19
  ASAT: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  ASAT: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  ASAT: SCR: Missing | 0 | 0 | 0 | 0 | 0
  ASAT: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ASAT: PRE: Below LLN | 0 | 0 | 0 | 0 | 1
  ASAT: PRE: Normal | 20 | 18 | 18 | 20 | 18
  ASAT: PRE: Grade 1-2 | 0 | 2 | 2 | 0 | 1
  ASAT: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  ASAT: PRE: Missing | 0 | 0 | 0 | 0 | 0
  ASAT: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ASAT: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  ASAT: PI(D7): Normal | 20 | 19 | 20 | 20 | 20
  ASAT: PI(D7): Grade 1-2 | 0 | 1 | 0 | 0 | 0
  ASAT: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  ASAT: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  ASAT: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ASAT: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 1
  ASAT: PI(D28): Normal | 19 | 19 | 20 | 19 | 18
  ASAT: PI(D28): Grade 1-2 | 1 | 0 | 0 | 0 | 1
  ASAT: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  ASAT: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  ASAT: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  ASAT: PII(D35): Below LLN | 0 | 1 | 1 | 0 | 0
  ASAT: PII(D35): Normal | 19 | 16 | 18 | 19 | 20
  ASAT: PII(D35): Grade 1-2 | 1 | 2 | 0 | 0 | 0
  ASAT: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  ASAT: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  ASAT: PII(D35): Grade 3 or more | 0 | 0 | 1 | 0 | 0
  ASAT: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  ASAT: PII(D56): Normal | 18 | 17 | 20 | 19 | 19
  ASAT: PII(D56): Grade 1-2 | 2 | 2 | 0 | 0 | 1
  ASAT: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  ASAT: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  ASAT: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  BUN: SCR: Below LLN | 0 | 1 | 0 | 1 | 0
  BUN: SCR: Normal | 20 | 19 | 20 | 19 | 20
  BUN: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  BUN: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  BUN: SCR: Missing | 0 | 0 | 0 | 0 | 0
  BUN: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  BUN: PRE: Below LLN | 1 | 1 | 0 | 1 | 0
  BUN: PRE: Normal | 19 | 19 | 20 | 19 | 20
  BUN: PRE: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  BUN: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  BUN: PRE: Missing | 0 | 0 | 0 | 0 | 0
  BUN: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  BUN: PI(D7): Below LLN | 0 | 1 | 1 | 1 | 0
  BUN: PI(D7): Normal | 20 | 19 | 19 | 19 | 20
  BUN: PI(D7): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  BUN: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  BUN: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  BUN: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  BUN: PI(D28): Below LLN | 1 | 0 | 0 | 0 | 0
  BUN: PI(D28): Normal | 19 | 19 | 20 | 19 | 20
  BUN: PI(D28): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  BUN: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  BUN: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  BUN: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  BUN: PII(D35): Below LLN | 0 | 1 | 1 | 1 | 0
  BUN: PII(D35): Normal | 20 | 18 | 19 | 18 | 20
  BUN: PII(D35): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  BUN: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  BUN: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  BUN: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  BUN: PII(D56): Below LLN | 0 | 0 | 0 | 1 | 1
  BUN: PII(D56): Normal | 20 | 19 | 20 | 18 | 19
  BUN: PII(D56): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  BUN: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  BUN: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  BUN: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Creatinine: SCR: Below LLN | 0 | 0 | 0 | 0 | 0
  Creatinine: SCR: Normal | 20 | 20 | 20 | 19 | 20
  Creatinine: SCR: Grade 1-2 | 0 | 0 | 0 | 1 | 0
  Creatinine: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Creatinine: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Creatinine: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Creatinine: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  Creatinine: PRE: Normal | 20 | 20 | 19 | 20 | 20
  Creatinine: PRE: Grade 1-2 | 0 | 0 | 1 | 0 | 0
  Creatinine: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  Creatinine: PRE: Missing | 0 | 0 | 0 | 0 | 0
  Creatinine: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D7): Normal | 20 | 19 | 19 | 20 | 20
  Creatinine: PI(D7): Grade 1-2 | 0 | 1 | 1 | 0 | 0
  Creatinine: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D28): Normal | 20 | 19 | 20 | 19 | 20
  Creatinine: PI(D28): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  Creatinine: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Creatinine: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D35): Below LLN | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D35): Normal | 20 | 19 | 20 | 19 | 19
  Creatinine: PII(D35): Grade 1-2 | 0 | 0 | 0 | 0 | 1
  Creatinine: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Creatinine: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D56): Normal | 20 | 19 | 20 | 19 | 20
  Creatinine: PII(D56): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  Creatinine: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Creatinine: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Eosinophils: SCR: Below LLN | 0 | 2 | 0 | 1 | 0
  Eosinophils: SCR: Normal | 20 | 17 | 20 | 19 | 20
  Eosinophils: SCR: Grade 1-2 | 0 | 1 | 0 | 0 | 0
  Eosinophils: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Eosinophils: PRE: Below LLN | 0 | 1 | 0 | 1 | 0
  Eosinophils: PRE: Normal | 20 | 18 | 20 | 18 | 20
  Eosinophils: PRE: Grade 1-2 | 0 | 1 | 0 | 1 | 0
  Eosinophils: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils: PRE: Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Eosinophils: PI(D7): Below LLN | 0 | 2 | 0 | 0 | 0
  Eosinophils: PI(D7): Normal | 20 | 17 | 19 | 19 | 20
  Eosinophils: PI(D7): Grade 1-2 | 0 | 1 | 1 | 1 | 0
  Eosinophils: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Eosinophils: PI(D28): Below LLN | 0 | 2 | 0 | 0 | 0
  Eosinophils: PI(D28): Normal | 20 | 17 | 18 | 19 | 20
  Eosinophils: PI(D28): Grade 1-2 | 0 | 0 | 2 | 0 | 0
  Eosinophils: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Eosinophils: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Eosinophils: PII(D35): Below LLN | 1 | 2 | 0 | 0 | 1
  Eosinophils: PII(D35): Normal | 19 | 17 | 19 | 19 | 19
  Eosinophils: PII(D35): Grade 1-2 | 0 | 0 | 1 | 0 | 0
  Eosinophils: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Eosinophils: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Eosinophils: PII(D56): Below LLN | 0 | 2 | 0 | 0 | 0
  Eosinophils: PII(D56): Normal | 19 | 17 | 19 | 18 | 20
  Eosinophils: PII(D56): Grade 1-2 | 1 | 0 | 1 | 1 | 0
  Eosinophils: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Eosinophils: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Hemoglobin: SCR: Below LLN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: SCR: Normal | 20 | 20 | 20 | 20 | 20
  Hemoglobin: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Hemoglobin: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PRE: Normal | 20 | 19 | 18 | 18 | 20
  Hemoglobin: PRE: Grade 1-2 | 0 | 1 | 2 | 2 | 0
  Hemoglobin: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PRE: Missing | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D7): Normal | 19 | 19 | 18 | 17 | 20
  Hemoglobin: PI(D7): Grade 1-2 | 1 | 1 | 2 | 3 | 0
  Hemoglobin: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D28): Normal | 20 | 17 | 18 | 16 | 20
  Hemoglobin: PI(D28): Grade 1-2 | 0 | 2 | 2 | 3 | 0
  Hemoglobin: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Hemoglobin: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PII(D35): Below LLN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PII(D35): Normal | 20 | 15 | 18 | 17 | 18
  Hemoglobin: PII(D35): Grade 1-2 | 0 | 4 | 2 | 2 | 2
  Hemoglobin: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Hemoglobin: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PII(D56): Normal | 20 | 16 | 19 | 17 | 20
  Hemoglobin: PII(D56): Grade 1-2 | 0 | 3 | 1 | 2 | 0
  Hemoglobin: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  Hemoglobin: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Hemoglobin: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Lymphocytes: SCR: Below LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: SCR: Normal | 20 | 20 | 20 | 20 | 20
  Lymphocytes: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PRE: Normal | 20 | 20 | 20 | 20 | 20
  Lymphocytes: PRE: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PRE: Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PI(D7): Normal | 20 | 19 | 20 | 20 | 20
  Lymphocytes: PI(D7): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PI(D7): Above ULN | 0 | 1 | 0 | 0 | 0
  Lymphocytes: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PI(D28): Normal | 20 | 18 | 20 | 18 | 19
  Lymphocytes: PI(D28): Grade 1-2 | 0 | 1 | 0 | 0 | 1
  Lymphocytes: PI(D28): Above ULN | 0 | 0 | 0 | 1 | 0
  Lymphocytes: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Lymphocytes: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D35): Below LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D35): Normal | 20 | 19 | 19 | 18 | 20
  Lymphocytes: PII(D35): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D35): Above ULN | 0 | 0 | 1 | 1 | 0
  Lymphocytes: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Lymphocytes: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D56): Normal | 20 | 19 | 20 | 19 | 20
  Lymphocytes: PII(D56): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  Lymphocytes: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Lymphocytes: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Neutrophils: SCR: Below LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils: SCR: Normal | 20 | 20 | 20 | 20 | 20
  Neutrophils: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Neutrophils: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Neutrophils: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Neutrophils: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils: PRE: Normal | 20 | 19 | 17 | 20 | 19
  Neutrophils: PRE: Grade 1-2 | 0 | 1 | 2 | 0 | 1
  Neutrophils: PRE: Above ULN | 0 | 0 | 1 | 0 | 0
  Neutrophils: PRE: Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Neutrophils: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils: PI(D7): Normal | 20 | 19 | 19 | 19 | 15
  Neutrophils: PI(D7): Grade 1-2 | 0 | 1 | 0 | 1 | 3
  Neutrophils: PI(D7): Above ULN | 0 | 0 | 1 | 0 | 2
  Neutrophils: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Neutrophils: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils: PI(D28): Normal | 20 | 19 | 18 | 19 | 20
  Neutrophils: PI(D28): Grade 1-2 | 0 | 0 | 1 | 0 | 0
  Neutrophils: PI(D28): Above ULN | 0 | 0 | 1 | 0 | 0
  Neutrophils: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Neutrophils: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Neutrophils: PII(D35): Below LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils: PII(D35): Normal | 19 | 18 | 20 | 19 | 17
  Neutrophils: PII(D35): Grade 1-2 | 0 | 1 | 0 | 0 | 0
  Neutrophils: PII(D35): Above ULN | 1 | 0 | 0 | 0 | 2
  Neutrophils: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Neutrophils: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 1
  Neutrophils: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils: PII(D56): Normal | 20 | 19 | 17 | 18 | 17
  Neutrophils: PII(D56): Grade 1-2 | 0 | 0 | 1 | 1 | 3
  Neutrophils: PII(D56): Above ULN | 0 | 0 | 2 | 0 | 0
  Neutrophils: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Neutrophils: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Platelets: SCR: Below LLN | 0 | 0 | 0 | 0 | 0
  Platelets: SCR: Normal | 20 | 20 | 20 | 20 | 20
  Platelets: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Platelets: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Platelets: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Platelets: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Platelets: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  Platelets: PRE: Normal | 19 | 20 | 19 | 20 | 19
  Platelets: PRE: Grade 1-2 | 1 | 0 | 1 | 0 | 1
  Platelets: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  Platelets: PRE: Missing | 0 | 0 | 0 | 0 | 0
  Platelets: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Platelets: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  Platelets: PI(D7): Normal | 20 | 20 | 20 | 20 | 19
  Platelets: PI(D7): Grade 1-2 | 0 | 0 | 0 | 0 | 1
  Platelets: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  Platelets: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Platelets: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Platelets: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  Platelets: PI(D28): Normal | 20 | 19 | 20 | 18 | 19
  Platelets: PI(D28): Grade 1-2 | 0 | 0 | 0 | 0 | 1
  Platelets: PI(D28): Above ULN | 0 | 0 | 0 | 1 | 0
  Platelets: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Platelets: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Platelets: PII(D35): Below LLN | 0 | 0 | 0 | 0 | 0
  Platelets: PII(D35): Normal | 20 | 19 | 20 | 18 | 20
  Platelets: PII(D35): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Platelets: PII(D35): Above ULN | 0 | 0 | 0 | 1 | 0
  Platelets: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Platelets: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Platelets: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  Platelets: PII(D56): Normal | 19 | 19 | 20 | 19 | 19
  Platelets: PII(D56): Grade 1-2 | 1 | 0 | 0 | 0 | 0
  Platelets: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 1
  Platelets: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Platelets: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  White blood cells: SCR: Below LLN | 0 | 0 | 0 | 0 | 0
  White blood cells: SCR: Normal | 20 | 17 | 20 | 20 | 18
  White blood cells: SCR: Grade 1-2 | 0 | 3 | 0 | 0 | 2
  White blood cells: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  White blood cells: SCR: Missing | 0 | 0 | 0 | 0 | 0
  White blood cells: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  White blood cells: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  White blood cells: PRE: Normal | 19 | 18 | 18 | 20 | 18
  White blood cells: PRE: Grade 1-2 | 1 | 2 | 2 | 0 | 2
  White blood cells: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  White blood cells: PRE: Missing | 0 | 0 | 0 | 0 | 0
  White blood cells: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D7): Normal | 19 | 18 | 17 | 19 | 15
  White blood cells: PI(D7): Grade 1-2 | 1 | 2 | 3 | 1 | 5
  White blood cells: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D28): Normal | 20 | 18 | 18 | 19 | 20
  White blood cells: PI(D28): Grade 1-2 | 0 | 1 | 2 | 0 | 0
  White blood cells: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  White blood cells: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  White blood cells: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  White blood cells: PII(D35): Below LLN | 0 | 0 | 0 | 0 | 0
  White blood cells: PII(D35): Normal | 18 | 16 | 19 | 19 | 17
  White blood cells: PII(D35): Grade 1-2 | 2 | 3 | 1 | 0 | 3
  White blood cells: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  White blood cells: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  White blood cells: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  White blood cells: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  White blood cells: PII(D56): Normal | 18 | 19 | 17 | 19 | 17
  White blood cells: PII(D56): Grade 1-2 | 2 | 0 | 3 | 0 | 3
  White blood cells: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  White blood cells: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  White blood cells: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Total bilibrubin: SCR: Below LLN | 0 | 0 | 0 | 1 | 0
  Total bilibrubin: SCR: Normal | 20 | 20 | 20 | 19 | 19
  Total bilibrubin: SCR: Grade 1-2 | 0 | 0 | 0 | 0 | 1
  Total bilibrubin: SCR: Above ULN | 0 | 0 | 0 | 0 | 0
  Total bilibrubin: SCR: Missing | 0 | 0 | 0 | 0 | 0
  Total bilibrubin: SCR: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PRE: Below LLN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PRE: Normal | 20 | 19 | 20 | 19 | 19
  Total bilirubin: PRE: Grade 1-2 | 0 | 0 | 0 | 1 | 1
  Total bilirubin: PRE: Above ULN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PRE: Missing | 0 | 1 | 0 | 0 | 0
  Total bilirubin: PRE: Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D7): Below LLN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D7): Normal | 20 | 20 | 20 | 20 | 20
  Total bilirubin: PI(D7): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D7): Above ULN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D7): Missing | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D7): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D28): Below LLN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D28): Normal | 20 | 19 | 20 | 19 | 19
  Total bilirubin: PI(D28): Grade 1-2 | 0 | 0 | 0 | 0 | 1
  Total bilirubin: PI(D28): Above ULN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PI(D28): Missing | 0 | 1 | 0 | 1 | 0
  Total bilirubin: PI(D28): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D35): Below LLN | 1 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D35): Normal | 19 | 19 | 20 | 19 | 20
  Total bilirubin: PII(D35): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D35): Above ULN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D35): Missing | 0 | 1 | 0 | 1 | 0
  Total bilirubin: PII(D35): Grade 3 or more | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D56): Below LLN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D56): Normal | 20 | 19 | 20 | 19 | 20
  Total bilirubin: PII(D56): Grade 1-2 | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D56): Above ULN | 0 | 0 | 0 | 0 | 0
  Total bilirubin: PII(D56): Missing | 0 | 1 | 0 | 1 | 0
  Total bilirubin: PII(D56): Grade 3 or more | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibody Titers Specific to Each DENV Type - According to Protocol Population (ATP)
Description: Geometric Mean Titers (GMTs) of Neutralizing antibody titers specific to each DENV type were measured by a quantitative microneutralization assay with a titer giving 50% reduction in viral infection (MN50) at specified time points. MN50 is specific and sensitive for the detection of anti-DENV neutralizing antibodies. The cut-off for seropositivity was 1: 10 for neutralizing antibody titers measured by MN50 assay. MN50 assay was used to determine initial DENV antibody status of subjects for inclusion in the ATP cohort.
  PRE = Pre-vaccination, Day 0 visit PI(D7) = Post-dose 1, Day 7 visit PI(D28) = Post-dose 1, Day 28 visit PII(D56) = Post-dose 2, Day 56 visit PII(M4) = Post-dose 2, Month 4 visit PII(M7) = Post-dose 2, Month 7 visit PII(M10) = Post-dose 2, Month 10 visit PII(M13) = Post-dose 2, Month 13 visit
Time Frame: up to month 13
Population: subjects with available data
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
GMT
  MN Ab Den1: PRE: number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den1: PRE | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PI(D7): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den1: PI(D7) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PI(D28): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den1: PI(D28) | 7.4 [5.5 to 10.1] | 16.7 [9.3 to 29.9] | 32.4 [14.8 to 71.0] | 28.9 [13.7 to 60.7] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PII(D56): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den1: PII(D56) | 64.3 [39.9 to 103.5] | 180.4 [122.6 to 265.4] | 335.8 [188.3 to 599.0] | 577.8 [340.3 to 981.4] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PII(M4): number analyzed (Participants) | 19 | 17 | 14 | 20 | 17
  MN Ab Den1: PII(M4) | 17.8 [9.5 to 33.4] | 129.6 [60.3 to 278.4] | 182.8 [90.7 to 368.7] | 247.6 [128.1 to 478.6] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PII(M7): number analyzed (Participants) | 18 | 17 | 12 | 16 | 17
  MN Ab Den1: PII(M7) | 7.2 [5.2 to 9.9] | 13.6 [8.9 to 20.8] | 21.5 [9.7 to 47.5] | 32.8 [18.6 to 57.8] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PII(M10): number analyzed (Participants) | 18 | 17 | 12 | 14 | 17
  MN Ab Den1: PII(M10) | 7.3 [4.9 to 10.8] | 14.5 [10.3 to 20.4] | 35.7 [11.9 to 106.9] | 24.3 [13.2 to 44.9] | 5.0 [5.0 to 5.0]
  MN Ab Den1: PII(M13): number analyzed (Participants) | 17 | 17 | 12 | 14 | 17
  MN Ab Den1: PII(M13) | 7.9 [5.3 to 12.0] | 13.2 [8.6 to 20.4] | 31.2 [9.6 to 101.2] | 24.9 [11.8 to 52.6] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PRE: number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den2: PRE | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PI(D7): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den2: PI(D7) | 5.0 [5.0 to 5.0] | 5.8 [4.2 to 8.2] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PI(D28): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den2: PI(D28) | 5.2 [4.8 to 5.7] | 18.1 [9.7 to 33.7] | 19.8 [8.2 to 48.0] | 15.9 [8.3 to 30.5] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PII(D56): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den2: PII(D56) | 44.2 [23.5 to 83.3] | 159.3 [96.2 to 263.8] | 361.4 [188.2 to 694.1] | 373.3 [194.7 to 715.6] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PII(M4): number analyzed (Participants) | 19 | 17 | 14 | 17 | 17
  MN Ab Den2: PII(M4) | 7.9 [5.7 to 10.8] | 23.1 [11.2 to 47.8] | 46.6 [23.4 to 93.0] | 47.2 [26.0 to 85.7] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PII(M7): number analyzed (Participants) | 18 | 17 | 12 | 16 | 17
  MN Ab Den2: PII(M7) | 5.9 [4.6 to 7.5] | 14.0 [8.5 to 23.2] | 19.9 [8.6 to 46.1] | 22.6 [12.3 to 41.5] | 5.0 [5.0 to 5.0]
  MN Ab Den2: PII(M10): number analyzed (Participants) | 18 | 17 | 12 | 14 | 17
  MN Ab Den2: PII(M10) | 6.4 [4.4 to 9.3] | 9.4 [5.5 to 16.0] | 43.6 [15.7 to 121.4] | 16.8 [9.1 to 31.0] | 5.0 [5.0 to 5.0]
  MN Ab Den: PII(M13): number analyzed (Participants) | 17 | 17 | 12 | 14 | 17
  MN Ab Den: PII(M13) | 7.2 [4.7 to 11.1] | 9.4 [6.0 to 14.6] | 27.3 [11.0 to 67.6] | 17.1 [8.6 to 34.0] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PRE: number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den3: PRE | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PI(D7): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den3: PI(D7) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PI(D28): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den3: PI(D28) | 5.3 [4.6 to 6.2] | 14.7 [8.3 to 26.0] | 20.0 [9.5 to 42.1] | 14.1 [6.8 to 29.4] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PII(D56): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den3: PII(D56) | 65.6 [41.1 to 104.8] | 188.9 [119.5 to 298.7] | 431.5 [222.0 to 838.7] | 495.5 [317.6 to 773.0] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PII(M4): number analyzed (Participants) | 19 | 17 | 14 | 17 | 17
  MN Ab Den3: PII(M4) | 13.2 [7.9 to 21.8] | 60.4 [35.8 to 101.7] | 135.4 [71.6 to 255.9] | 129.6 [68.0 to 246.8] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PII(M7): number analyzed (Participants) | 18 | 17 | 12 | 16 | 17
  MN Ab Den3: PII(M7) | 5.8 [4.7 to 7.1] | 13.4 [9.4 to 19.2] | 21.0 [9.6 to 46.0] | 29.5 [13.8 to 62.8] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PII(M10): number analyzed (Participants) | 18 | 17 | 12 | 14 | 17
  MN Ab Den3: PII(M10) | 6.0 [4.6 to 7.8] | 9.1 [6.0 to 13.9] | 36.7 [12.4 to 108.9] | 20.7 [10.7 to 40.1] | 5.0 [5.0 to 5.0]
  MN Ab Den3: PII(M13): number analyzed (Participants) | 17 | 17 | 12 | 14 | 17
  MN Ab Den3: PII(M13) | 5.7 [4.6 to 7.1] | 9.5 [6.1 to 14.7] | 36.7 [14.9 to 90.8] | 24.0 [11.6 to 49.8] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PRE: number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den4: PRE | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PI(D7): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den4: PI(D7) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PI(D28): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den4: PI(D28) | 5.3 [4.6 to 6.2] | 8.2 [4.1 to 16.4] | 6.7 [4.3 to 10.6] | 7.4 [4.1 to 13.2] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PII(D56): number analyzed (Participants) | 19 | 17 | 14 | 17 | 18
  MN Ab Den4: PII(D56) | 26.0 [10.8 to 62.3] | 162.7 [67.0 to 394.9] | 201.7 [66.2 to 614.8] | 462.3 [217.6 to 981.9] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PII(M4): number analyzed (Participants) | 19 | 17 | 14 | 17 | 17
  MN Ab Den4: PII(M4) | 5.9 [4.9 to 7.2] | 12.9 [7.2 to 23.0] | 17.6 [7.5 to 41.2] | 29.8 [13.4 to 66.2] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PII(M7): number analyzed (Participants) | 18 | 17 | 12 | 16 | 17
  MN Ab Den4: PII(M7) | 6.0 [4.8 to 7.5] | 9.1 [5.2 to 15.8] | 7.5 [3.8 to 15.0] | 15.2 [6.7 to 34.6] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PII(M10): number analyzed (Participants) | 18 | 17 | 12 | 14 | 17
  MN Ab Den4: PII(M10) | 5.8 [4.7 to 7.1] | 7.1 [4.6 to 11.0] | 11.0 [4.4 to 27.1] | 6.8 [4.6 to 10.0] | 5.0 [5.0 to 5.0]
  MN Ab Den4: PII(M13): number analyzed (Participants) | 17 | 17 | 12 | 14 | 17
  MN Ab Den4: PII(M13) | 5.3 [4.7 to 6.1] | 7.3 [4.2 to 12.8] | 9.3 [3.9 to 22.2] | 8.2 [4.7 to 14.3] | 5.0 [5.0 to 5.0]

8. Secondary Outcome: Number of Subject Showing Monovalent, Bivalent, Trivalent and Tetravalent Response for Neutralizing Antibodies - Total Vaccinated Cohort (TVC)
Description: Number of subjects showing Monovalent, bivalent, trivalent and tetravalent response for neutralizing antibodies by Microneutralization Titer (giving 50% reduction in viral infection (MN50)) in the TVC population.
  PI(D7) = Post-dose 1, Day 7 visit PI(D28) = Post-dose 1, Day 28 visit PII(D56) = Post-dose 2, Day 56 visit PII(M4) = Post-dose 2, Month 4 visit PII(M7) = Post-dose 2, Month 7 visit PII(M10) = Post-dose 2, Month 10 visit PII(M13) = Post-dose 2, Month 13 visit
Time Frame: up to month 13
Population: subjects with available results for all four DENV-types (without missing N antibody titer)
Measure: Count of Participants; unit: Participants
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Participants
  PRE: None | 20 | 19 | 16 | 19 | 18
  PRE: Monovalent | 0 | 0 | 2 | 0 | 0
  PRE: Bivalent | 0 | 0 | 0 | 0 | 0
  PRE: Trivalent | 0 | 0 | 2 | 0 | 0
  PRE: Tetravalent | 0 | 1 | 0 | 1 | 2
  PI(D7): None | 20 | 18 | 16 | 19 | 18
  PI(D7): Monovalent | 0 | 1 | 1 | 0 | 0
  PI(D7): Bivalent | 0 | 0 | 1 | 0 | 0
  PI(D7): Trivalent | 0 | 0 | 1 | 0 | 0
  PI(D7): Tetravalent | 0 | 1 | 1 | 1 | 2
  PI(D28): number analyzed (Participants) | 20 | 19 | 20 | 19 | 20
  PI(D28): None | 14 | 3 | 2 | 4 | 18
  PI(D28): Monovalent | 4 | 3 | 5 | 3 | 0
  PI(D28): Bivalent | 1 | 4 | 2 | 4 | 0
  PI(D28): Trivalent | 1 | 5 | 6 | 5 | 0
  PI(D28): Tetravalent | 0 | 4 | 5 | 3 | 2
  PII(56): number analyzed (Participants) | 20 | 19 | 20 | 19 | 20
  PII(56): None | 0 | 0 | 0 | 0 | 18
  PII(56): Monovalent | 0 | 0 | 0 | 0 | 0
  PII(56): Bivalent | 1 | 0 | 0 | 0 | 0
  PII(56): Trivalent | 7 | 1 | 1 | 0 | 0
  PII(56): Tetravalent | 12 | 18 | 19 | 19 | 2
  PII(M4): number analyzed (Participants) | 20 | 18 | 20 | 19 | 19
  PII(M4): None | 5 | 0 | 0 | 0 | 17
  PII(M4): Monovalent | 6 | 0 | 0 | 0 | 0
  PII(M4): Bivalent | 2 | 5 | 2 | 2 | 0
  PII(M4): Trivalent | 4 | 3 | 7 | 3 | 0
  PII(M4): Tetravalent | 3 | 10 | 11 | 14 | 2
  PII(M7): number analyzed (Participants) | 19 | 18 | 18 | 18 | 19
  PII(M7): None | 12 | 2 | 1 | 2 | 17
  PII(M7): Monovalent | 5 | 2 | 3 | 1 | 0
  PII(M7): Bivalent | 0 | 4 | 3 | 3 | 0
  PII(M7): Trivalent | 1 | 4 | 6 | 5 | 0
  PII(M7): Tetravalent | 1 | 6 | 5 | 7 | 2
  PII(M10): number analyzed (Participants) | 19 | 18 | 19 | 16 | 19
  PII(M10): None | 15 | 3 | 0 | 2 | 17
  PII(M10): Monovalent | 2 | 6 | 4 | 2 | 0
  PII(M10): Bivalent | 0 | 2 | 4 | 1 | 0
  PII(M10): Trivalent | 0 | 3 | 3 | 7 | 0
  PII(M10): Tetravalent | 2 | 4 | 8 | 4 | 2
  PII(M13): number analyzed (Participants) | 18 | 18 | 19 | 16 | 19
  PII(M13): None | 12 | 5 | 2 | 3 | 17
  PII(M13): Monovalent | 4 | 4 | 1 | 2 | 0
  PII(M13): Bivalent | 0 | 3 | 5 | 0 | 0
  PII(M13): Trivalent | 1 | 2 | 5 | 6 | 0
  PII(M13): Tetravalent | 1 | 4 | 6 | 5 | 2

ADVERSE EVENTS:
Time Frame: days 0-392
Arm/Group | TDENV-PIV alum1 | TDENV-PIV alum4 | TDENV-PIV AS01E1 | TDENV-PIV AS03B1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 1/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20 | 3/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 9/20 | 12/20 | 15/20 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDENV-PIV alum1 (N=20) | TDENV-PIV alum4 (N=20) | TDENV-PIV AS01E1 (N=20) | TDENV-PIV AS03B1 (N=20) | Placebo (N=20)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miscarriage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gunshot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDENV-PIV alum1 (N=20) | TDENV-PIV alum4 (N=20) | TDENV-PIV AS01E1 (N=20) | TDENV-PIV AS03B1 (N=20) | Placebo (N=20)
Ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bacterial vaginosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bruise at injection site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash on chest (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Contact dermatitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased heart rate (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Decreased hemoglobin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Decreased neutrophils (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 3 (4)
Decreased platelets (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Direct bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated creatinine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated ALT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated AST (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated heart rate (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Elevated systolic blood pressure (Investigations) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Elevated WBC (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Forgetfulness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gunshot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Increased heart rate (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased WBC (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left arm fell asleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Miscarriage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle soreness, back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain, left side (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmares (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain from skin abrasion, left knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain, ear piercing (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain, groin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right upper thigh pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tenderness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Strep throat (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sweats (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope vasovagal (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 3 (6) | 2 (2)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening uterin fibroids (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No